CLINICAL TRIAL: NCT01591733
Title: Phase II Study of Preoperative FOLFIRINOX Followed by Accelerated Short Course Radiation Therapy for Borderline-Resectable Pancreatic Cancer
Brief Title: FOLFIRINOX + RT for Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Theodore Sunki Hong, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-328
Record Dates: First submitted 2012-04-20; First posted 2012-05-04 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Cancer
Keywords: Borderline resectable
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox; Fluorouracil; Oxaliplatin; Irinotecan; Capecitabine; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): All participants will receive the FOLFIRINOX regimen, followed by capecitabine and short course radiation therapy.
  Interventions: Drug: FOLFIRINOX; Drug: Capecitabine; Radiation: Short Course Radiation; Procedure: Surgery

INTERVENTIONS:
Drug: FOLFIRINOX — Up to Eight-14 day cycles
  Other Names: 5-FU; Oxaliplatin; Irinotecan
Drug: Capecitabine — Orally, for 10 days
Radiation: Short Course Radiation — Five or ten days
Procedure: Surgery — 1-4 weeks after completion of capecitabine therapy

SUMMARY:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of a therapy to learn whether the therapy works in treating a specific cancer. "Investigational" means that the therapy is still being studied and that research doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause, and if therapy is effective for treating different types of cancer. Proton beam radiation therapy is an FDA (U.S. Food and Drug Administration) approved radiation delivery system.

Proton beam radiation therapy is known to spare surrounding normal tissues from radiation as it delivers less radiation beyond the area of the target tissues. This may reduce side effects that patients would normally experience with standard (photon) radiation therapy, which tends to include more normal tissue along with tumor target tissue.

Researchers in the laboratory have discovered that there are pathways inside the cells that can lead to growth and survival of the tumor. The chemotherapy drugs FOLFIRINOX and capecitabine are targeted towards blocking the pathways that allow cancer cells to divide, and may result in the tumor shrinking in size.

In this research study, the investigators are looking to determine if proton beam radiation in combination with FOLFIRINOX and capecitabine is effective in controlling the growth of your cancer.

DETAILED DESCRIPTION:
For weeks 1-8, you will only be receiving FOLFIRINOX via IV infusion. The treatment plan will begin with four cycles (8 weeks) of FOLFIRINOX. Each cycle is 14 days long. You will receive FOLFIRINOX therapy on days 1, 2 and 3 of each of the four cycles. The FOLFIRINOX treatment is broken up into three different drugs. 5-FU will be administered over two hours on day one of each cycle, and then continuously with a pump for days 2 and 3. Oxaliplatin will be delivered by intravenous (infusion) over 120 minutes. Irinotecan will be given by IV for 90 minutes. All parts of this treatment will be received as an outpatient.

If after 4 cycles of FOLFIRINOX therapy, your tumor has not spread, you will receive a further 4 cycles of FOLFIRINOX. If after 8 total cycles of FOLFIRINOX your cancer is clearly resectable, you will proceed to phase 2 of treatment with capecitabine and radiation therapy.

You will take tablets of capecitabine by mouth for a total of 10 days (Monday through Friday) during the two weeks after your FOLFIRINOX treatment.

You will be given a drug diary for capecitabine which contains instructions on how to take the drug.

Short course radiation: You will receive proton radiation treatment for five days (Monday through Friday) after your FOLFIRINOX treatment, during the time of your capecitabine treatment, or photon radiation for ten days (Monday through Friday for two weeks). You will also be assessed at least once during this treatment course for any side effects you may be experiencing.

You will receive study radiation treatment as an outpatient at the Francis H. Burr Proton Center or the Clark Center for Radiation Oncology at the Massachusetts General Hospital Surgery is expected to occur approximately one to four weeks after completion of capecitabine therapy.

After your surgery, you may receive additional chemotherapy at the discretion of your treating physician and be followed as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic proof pancreatic ductal carcinoma
* Borderline resectable
* Life expectancy of at least 3 months
* ECOG Performance Status ≤ 1
* Adequate organ and bone marrow function
* No treatment of other invasive cancers within the last 5 years with greater than 5% risk of recurrence at the time of eligibility screening. Carcinoma in-situ and basal cell carcinoma/squamous cell carcinoma of the skin are allowed
* > 4 weeks since major surgery, excluding laparoscopy

Exclusion Criteria:

* Evidence of metastatic disease
* Pregnant or breastfeeding
* Other serious uncontrolled medical conditions
* Prior chemotherapy, targeted/biologic therapy or radiation for treatment of the pancreatic tumor
* Prior systemic fluoropyrimidine therapy
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability
* Individuals on cimetidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2022-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S Hong, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Murphy JE, Wo JY, Ryan DP, Jiang W, Yeap BY, Drapek LC, Blaszkowsky LS, Kwak EL, Allen JN, Clark JW, Faris JE, Zhu AX, Goyal L, Lillemoe KD, DeLaney TF, Fernandez-Del Castillo C, Ferrone CR, Hong TS. Total Neoadjuvant Therapy With FOLFIRINOX Followed by Individualized Chemoradiotherapy for Borderline Resectable Pancreatic Adenocarcinoma: A Phase 2 Clinical Trial. JAMA Oncol. 2018 Jul 1;4(7):963-969. doi: 10.1001/jamaoncol.2018.0329. PMID 29800971

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFIRINOX + Radiation: All participants will receive the FOLFIRINOX regimen, followed by capecitabine and short course radiation therapy.
  FOLFIRINOX: Up to Eight-14 day cycles
  Capecitabine: Orally, for 10 days
  Short Course Radiation: Five or ten days
  Surgery: 1-4 weeks after completion of capecitabine therapy
Period: Overall Study
Arm/Group | FOLFIRINOX + Radiation
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FOLFIRINOX + Radiation
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 62 [46 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48
CA19-9 Level [Count of Participants; unit: Participants] — Cancer antigen 19-9 (CA 19-9) level
  Participants
    <35 U/ml (Normal) | 12
    ≥35 U/ml (elevated) | 36
CEA Level [Count of Participants; unit: Participants] — Carcinoembryonic antigen level
  Participants
    <3.4 ng/ml (normal) | 23
    ≥3.4 ng/ml (elevated) | 25
Pancreatic Tumor Site [Count of Participants; unit: Participants]
  Head | 35
  Body | 11
  Tail | 2
Tumor Size [Median (Full Range); unit: Centimeters (cm)] | 3.75 [2.1 to 5.6]
Vessel Involvement [Count of Participants; unit: Participants]
  Venous | 28
  Arterial | 7
  Both | 12
  None | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of R0 Resection
Description: The rate of R0 resection of patients with borderline-resectable adenocarcinoma of the head of the pancreas, along with borderline-resectable and resectable adenocarcinoma of the body and tail of the pancreas. R0 resection means that following surgery, no cancer cells are seen microscopically at the resection margin.
Time Frame: Post-surgery (about 4 months post baseline)
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible - FOLFIRINOX + Radiation: The overall study population
  All participants will receive the FOLFIRINOX regimen, followed by capecitabine and short course radiation therapy.
  FOLFIRINOX: Up to Eight-14 day cycles
  Capecitabine: Orally, for 10 days
  Short Course Radiation: Five or ten days
  Surgery: 1-4 weeks after completion of capecitabine therapy
- Resected Participants - FOLFIRINOX + Radiation: The participants that were resected.
  All participants will receive the FOLFIRINOX regimen, followed by capecitabine and short course radiation therapy.
  FOLFIRINOX: Up to Eight-14 day cycles
  Capecitabine: Orally, for 10 days
  Short Course Radiation: Five or ten days
  Surgery: 1-4 weeks after completion of capecitabine therapy
Arm/Group | All Eligible - FOLFIRINOX + Radiation | Resected Participants - FOLFIRINOX + Radiation
Number analyzed (Participants) | 48 | 32
Participants | 31 | 31

2. Secondary Outcome: Median Progression-Free Survival
Description: The median progression free survival as measured from the start of treatment until the time of disease progression or death, whichever occurs first. Disease status was evaluated using RECIST (Response Evaluation Criteria in Solid Tumors). Disease progression is defined as having at least a 20% increase in the sum of the longest diameter (LD) of target lesion, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From the start of treatment until death or disease progression, median duration of follow-up of 14.7 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FOLFIRINOX + Radiation
Number analyzed (Participants) | 48
Months | 14.7 [10.5 to NA] — Upper bound is not defined due to skewed survival data (participants still surviving).

3. Secondary Outcome: Median Overall Survival
Description: Median overall survival, as measured from the start of treatment until the time of death.
Time Frame: From the start of treatment until the time of death, median duration of follow-up of 37.7 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FOLFIRINOX + Radiation
Number analyzed (Participants) | 48
Months | 37.7 [19.4 to NA] — Upper bound is not defined due to skewed survival data (participants still surviving).

4. Secondary Outcome: Preoperative Toxicity of Grade 3 or Worse Related to FOLFIRINOX and Chemoradiation
Description: Frequency of grade 3 or greater adverse events deemed related to FOLFIRINOX+short course radiation therapy. Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE 4).
Time Frame: From the start of treatment until the end of chemoradiation, about 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRINOX + Radiation
Number analyzed (Participants) | 48
Participants
  Diarrhea | 5
  Neutropenia | 2
  Febrile neutropenia | 1
  Lymphopenia | 1
  Thrombocytopenia | 1
  Anemia | 1
  Elevated alkaline phosphatase | 1
  Elevated bilirubin | 1
  Elevated AST/ALT | 1
  Peripheral neuropathy | 2
  Abdominal pain | 1
  Constipation | 1

5. Secondary Outcome: The Proportion of Participants With Surgery Related Adverse Events
Description: The number of participants with surgery related any grade adverse events following pancreaticoduodenectomy or distal pancreatectomy after receiving preoperative FOLFIRINOX and preoperative short course radiation therapy. Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE 4).
Time Frame: At the time of surgery, 30 days post-surgery
Population: The participants that underwent surgery
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | FOLFIRINOX + Radiation
Number analyzed (Participants) | 32
proportion of participants | 0.375 [0.233 to 0.536]

6. Secondary Outcome: 30 Day Post-operative Mortality Rate
Description: The number of participants that died within 30 days after undergoing pancreaticoduodenectomy or distal pancreatectomy.
Time Frame: 30 days post surgery (about 6 months from baseline)
Population: The number of participants that underwent surgery
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRINOX + Radiation
Number analyzed (Participants) | 32
Participants | 0

7. Secondary Outcome: Rate of Pathologic Downstaging
Description: To determine the rate of pathologic down-staging among participants that underwent pancreaticoduodenectomy or distal pancreatectomy. The pathologic downstaging rate is the proportion of patients with the primary tumor and nodes downstaged based on final pathology of the surgical specimen.
Time Frame: Baseline, Post surgery
Reporting Status: Not Posted, anticipated posting 2022-01

8. Secondary Outcome: Local Control Rates
Description: The number of participants that achieved local control. Local control was evaluated using RECIST (Response Evaluation Criteria in Solid Tumors). Local Failure is defined as progression of the primary tumor, or to the reappearance of tumor at the primary site.
Time Frame: From the start of treatment until the end of treatment with FOLFIRINOX, or until disease progression (median duration of follow-up of approximately 14 months)
Population: The first 5 participants treated who only received 4 cycles of FOLFIRINOX instead of 8 were not included in the analysis of local control.
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRINOX + Radiation
Number analyzed (Participants) | 43
Participants | 32

9. Secondary Outcome: Correlation of Mutational Analysis Biomarkers
Description: To correlate mutational analysis biomarkers (SNaPSHOT assay) with response to treatment
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2022-01

10. Secondary Outcome: Quality of Life, Symptom Burden, and Mood
Description: Patient-reported outcomes: We will use descriptive statistics to describe Quality of Life (QOL) (EORTC QLQ-C30), symptom burden (ESAS-r) and mood (HADS) for the entire study cohort.
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2022-01

11. Secondary Outcome: Utilization of Health Services (Emergency Room, Hospital and Intensive Care Unit)
Description: Summary of the number of hospitalizations, intensive care unit (ICU) stays, emergency department (ED) stays, and palliative care use for the study population.
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2022-01

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of treatment, about 6 months. Treatment is continued until disease progression, intercurrent illness that prevents further treatment, unacceptable adverse events, participant withdrawal, or until the treating investigator decides it is in the participants best interest.
Description: Adverse events were defined as any grade 3 or greater toxicity deemed to be possibly, probably, or definitely related to treatment
Arm/Group | FOLFIRINOX + Radiation
All-Cause Mortality (participants affected / at risk) | 2/48
Serious Adverse Events (participants affected / at risk) | 24/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRINOX + Radiation (N=48)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (4)
Alkaline phosphatase increased (Investigations) | 2 (4)
Anaphylaxis (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Blood bilirubin increased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (11)
Fatigue (General disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4)
Fever (General disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 7 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Platelet count decreased (Investigations) | 2 (4)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRINOX + Radiation (N=48)
Abdominal distension (Gastrointestinal disorders) | 18 (38)
Abdominal pain (Gastrointestinal disorders) | 44 (187)
Alanine aminotransferase increased (Investigations) | 20 (43)
Alkaline phosphatase increased (Investigations) | 6 (12)
Allergic reaction (Immune system disorders) | 4 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (55)
Anemia (Blood and lymphatic system disorders) | 7 (14)
Anorexia (Metabolism and nutrition disorders) | 45 (163)
Anxiety (Psychiatric disorders) | 26 (70)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (17)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Ascites (Gastrointestinal disorders) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 10 (33)
Atrial fibrillation (Cardiac disorders) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (72)
Biliary tract infection (Infections and infestations) | 6 (7)
Bloating (Gastrointestinal disorders) | 16 (33)
Blood bilirubin increased (Investigations) | 16 (31)
Blurred vision (Eye disorders) | 5 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 12 (22)
Bruising (Injury, poisoning and procedural complications) | 10 (15)
Cardiac disorders - Other (Cardiac disorders) | 9 (17)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6 (8)
Chills (General disorders) | 16 (21)
Cholesterol high (Investigations) | 4 (4)
Cognitive disturbance (Nervous system disorders) | 3 (3)
Concentration impairment (Nervous system disorders) | 3 (4)
Confusion (Psychiatric disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 40 (114)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (34)
Dehydration (Metabolism and nutrition disorders) | 25 (69)
Depression (Psychiatric disorders) | 15 (28)
Diarrhea (Gastrointestinal disorders) | 43 (201)
Dizziness (Nervous system disorders) | 24 (55)
Dry eye (Eye disorders) | 3 (6)
Dry mouth (Gastrointestinal disorders) | 11 (15)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (16)
Dysarthria (Nervous system disorders) | 5 (9)
Dysesthesia (Nervous system disorders) | 3 (4)
Dysgeusia (Nervous system disorders) | 25 (36)
Dyspepsia (Gastrointestinal disorders) | 12 (20)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (33)
Edema face (General disorders) | 4 (4)
Edema limbs (General disorders) | 18 (51)
Enterocolitis (Gastrointestinal disorders) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (19)
Eye disorders - Other (Eye disorders) | 7 (11)
Eye pain (Eye disorders) | 3 (6)
Facial pain (General disorders) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 5 (7)
Fatigue (General disorders) | 48 (258)
Fecal incontinence (Gastrointestinal disorders) | 5 (7)
Fever (General disorders) | 28 (44)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 20 (57)
Flushing (Vascular disorders) | 3 (4)
Gait disturbance (General disorders) | 8 (14)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 17 (28)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 26 (54)
Gastroparesis (Gastrointestinal disorders) | 4 (8)
General disorders and administration site conditions - Other (General disorders) | 11 (39)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9 (28)
Hallucinations (Psychiatric disorders) | 3 (4)
Headache (Nervous system disorders) | 14 (31)
Hemorrhoids (Gastrointestinal disorders) | 4 (5)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 10 (28)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (6)
Hypertension (Vascular disorders) | 13 (19)
Hypokalemia (Metabolism and nutrition disorders) | 20 (92)
Hyponatremia (Metabolism and nutrition disorders) | 7 (9)
Hypotension (Vascular disorders) | 16 (26)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Infections and infestations - Other (Infections and infestations) | 10 (16)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 4 (4)
Insomnia (Psychiatric disorders) | 32 (78)
Lethargy (Nervous system disorders) | 3 (3)
Malabsorption (Gastrointestinal disorders) | 13 (20)
Malaise (General disorders) | 7 (13)
Memory impairment (Nervous system disorders) | 4 (4)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 4 (4)
Mucosal infection (Infections and infestations) | 3 (5)
Mucositis oral (Gastrointestinal disorders) | 20 (36)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 8 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (18)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Nausea (Gastrointestinal disorders) | 46 (217)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (7)
Nervous system disorders - Other (Nervous system disorders) | 7 (13)
Neutrophil count decreased (Investigations) | 6 (10)
Non-cardiac chest pain (General disorders) | 5 (9)
Oral pain (Gastrointestinal disorders) | 3 (3)
Pain (General disorders) | 7 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (18)
Pain of skin (Skin and subcutaneous tissue disorders) | 4 (4)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 (8)
Palpitations (Cardiac disorders) | 6 (9)
Pancreatic enzymes decreased (Investigations) | 6 (11)
Pancreatitis (Gastrointestinal disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 9 (14)
Peripheral motor neuropathy (Nervous system disorders) | 4 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 46 (243)
Platelet count decreased (Investigations) | 11 (21)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (14)
Rectal pain (Gastrointestinal disorders) | 3 (7)
Renal and urinary disorders - Other (Renal and urinary disorders) | 5 (7)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 3 (4)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 11 (15)
Sepsis (Infections and infestations) | 3 (4)
Sinus tachycardia (Cardiac disorders) | 7 (8)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 23 (51)
Skin infection (Infections and infestations) | 5 (7)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Somnolence (Nervous system disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 9 (18)
Spasticity (Nervous system disorders) | 8 (19)
Supraventricular tachycardia (Cardiac disorders) | 4 (4)
Thromboembolic event (Vascular disorders) | 5 (5)
Toothache (Gastrointestinal disorders) | 3 (4)
Tremor (Nervous system disorders) | 3 (7)
Upper respiratory infection (Infections and infestations) | 8 (11)
Urinary frequency (Renal and urinary disorders) | 10 (20)
Urinary incontinence (Renal and urinary disorders) | 4 (8)
Urinary tract infection (Infections and infestations) | 7 (16)
Urinary tract pain (Renal and urinary disorders) | 3 (5)
Urinary urgency (Renal and urinary disorders) | 5 (6)
Urine discoloration (Renal and urinary disorders) | 8 (12)
Vomiting (Gastrointestinal disorders) | 30 (73)
Watering eyes (Eye disorders) | 3 (5)
Weight gain (Investigations) | 3 (5)
Weight loss (Investigations) | 41 (163)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Wound complication (Injury, poisoning and procedural complications) | 3 (5)
Wound dehiscence (Injury, poisoning and procedural complications) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT01591733/Prot_SAP_000.pdf